CLINICAL TRIAL: NCT00159783
Title: A Double-Blind, 40-Week Continuation Study Evaluating the Safety of Asenapine and Olanzapine in the Treatment of Subjects With Acute Mania Clinical Trial Protocol A7501007 (Secondary Title: ARES)
Brief Title: 40 Week Extension Study Of Asenapine and Olanzapine For Bipolar Disorder (A7501007)(COMPLETED)(P05857)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05857; A7501007
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2010-07-16 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asenapine (Experimental): Asenapine 5-10 mg twice daily for 40 weeks
  Interventions: Drug: asenapine
- Olanzapine (Active Comparator): Olanzapine 5-20 mg once daily for 40 weeks
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: asenapine — Asenapine, 40 weeks
  Other Names: Org 5222
  Arms: Asenapine
Drug: Olanzapine — Olanzapine, 40 weeks
  Arms: Olanzapine

SUMMARY:
Bipolar disorder is characterized by mood swings that range from from high (manic) to low (depressed) states. Sometimes, symptoms of both depression and mania are present (mixed episodes). Asenapine is an investigational medication for the treatment of manic or mixed episodes of bipolar disorder. Patients who completed study A7501006 (a 9 week extension study) could continue with the same treatment that they had been receiving: asenapine or olanzapine (a medication that is already approved for the treatment of bipolar mania) in a 40 -week continuation study.

ELIGIBILITY:
Inclusion Criteria:

* Have completed asenapine 3-week and 9 -week studies for the treatment of an acute manic or mixed episode and not had any major protocol violations..

Exclusion Criteria:

* Patients with unstable medical conditions or clinically significant laboratory

abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2005-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

REFERENCES:
- [Result] McIntyre RS, Cohen M, Zhao J, Alphs L, Macek TA, Panagides J. Asenapine for long-term treatment of bipolar disorder: a double-blind 40-week extension study. J Affect Disord. 2010 Nov;126(3):358-65. doi: 10.1016/j.jad.2010.04.005. PMID 20537396

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Asenapine: Asenapine 5-10 mg twice daily for 40 weeks (participants who were on placebo during the 3 week core study)
- Asenapine: Asenapine 5-10 mg twice daily for 40 weeks (participants who were on asenapine in the 3 week core study)
Period: Overall Study
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Started | 32 | 79 | 107
Completed | 13 | 52 | 68
Not Completed | 19 | 27 | 39
Not completed — Adverse Event | 5 | 7 | 9
Not completed — Lack of Efficacy | 1 | 2 | 3
Not completed — Withdrawal by Subject | 7 | 11 | 12
Not completed — Lost to Follow-up | 6 | 5 | 11
Not completed — Other | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine | Total
Number analyzed (Participants) | 32 | 79 | 107 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 77 | 106 | 214
  >=65 years | 1 | 2 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 43 | 39 | 97
  Male | 17 | 36 | 68 | 121

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Experienced Adverse Event(s)
Description: Adverse event (AE) data, both serious and non-serious, were collected. Serious AEs were also collected up to 30 days post last dose of study drug.
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product. It does not necessarily have to have a causal relationship with this treatment.
  An AE is defined as serious if it results in death, is life-threatening, requires in-patient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Up to 40 weeks
Measure: Number; unit: Participants
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Number analyzed (Participants) | 32 | 79 | 107
Participants | 23 | 68 | 85

2. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical exam (PE) included assessment of general appearance, skin, head, eyes, ears, nose, throat, lungs, blood pressure, cardiac rhythm & rate, neurologic status, and abdomen. The findings were deemed to be normal/abnormal based on the clinical judgment of the investigator.
Time Frame: Week 40 or endpoint
Measure: Number; unit: Participants
Groups:
- All Treatment Groups: Asenapine 5-10 mg twice daily for 40 weeks or Olanzapine 5-20 mg daily for 40 weeks
Arm/Group | All Treatment Groups
Number analyzed (Participants) | 218
Participants | 32

3. Primary Outcome: Number of Participants With Abnormal Electrocardiogram
Description: This is the number of participants with electrocardiogram (ECG) adverse events.
Time Frame: Week 40 or endpoint
Measure: Number; unit: Participants
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Number analyzed (Participants) | 32 | 79 | 107
Participants
  Sinus bradycardia | 0 | 2 | 0
  Bundle branch block right | 0 | 1 | 0
  ECG QRS complex prolonged | 0 | 0 | 1
  ECG ST segment depression | 0 | 0 | 1
  ECG T wave inversion | 0 | 0 | 1
  Supraventricular extrasystoles | 0 | 0 | 1
  Ventricular extrasystoles | 0 | 0 | 1

4. Primary Outcome: Body Weight
Description: Weight change from baseline
Time Frame: Baseline to Week 40 or endpoint
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Number analyzed (Participants) | 32 | 79 | 107
Kilograms
  Baseline | 81.4 (19.94) | 68.1 (17.22) | 72.0 (19.96)
  Change from baseline to Week 40 or endpoint | 1.7 (5.95) | 3.5 (6.65) | 6.0 (6.59)

5. Primary Outcome: Extrapyramidal Symptoms [EPS]
Description: EPS was assessed using the (1) involuntary movement scale [AIMS], (2) Barnes Akathisia Rating Scale [BARS], and (3) Simpson Angus Rating Scale SARS.
  AIMS score range 0-4; higher scores indicate greater symptom severity.
  BARS score rang 0-9; higher scores indicate greater severity of akathisia.
  SARS score range 0-40; higher scores indicate greater degree of Parkinsonism.
Time Frame: Week 40 or endpoint
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Number analyzed (Participants) | 32 | 79 | 107
Units on a scale
  AIMS | 0.4 (1.37) | 0.1 (0.60) | 0.0 (0.14)
  BARS | 0.4 (1.21) | 0.2 (0.77) | 0.1 (0.55)
  SARS | 0.6 (1.72) | 0.2 (1.36) | 0.3 (1.15)

6. Primary Outcome: Concomitant Medications
Description: Concomitant medications are any medications taken on or after the date of first dose of double-blind study drug through the date of
  last dose of double-blind study drug.
Time Frame: Up to 40 weeks
Measure: Number; unit: Participants
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Number analyzed (Participants) | 32 | 79 | 107
Participants
  Participants with no concomitant medications | 10 | 21 | 31
  Participants with >=1 concomitant medication | 22 | 58 | 76

7. Primary Outcome: Abdominal Girth
Description: Change in abdominal girth from baseline
Time Frame: Baseline to Week 40 or endpoint
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Number analyzed (Participants) | 32 | 79 | 107
Centimeters (cm)
  Baseline | 91.1 (14.20) | 86.8 (14.79) | 89.4 (14.78)
  Change from baseline to Week 40 or endpoint | 3.0 (6.84) | 2.6 (6.87) | 5.0 (7.89)

8. Primary Outcome: Number of Participants With Markedly Abnormal Vital Sign Changes
Description: Vital signs measured: sitting blood pressure, heart rate.
  Definitions:
  Markedly abnormal decreases: heart rate (HR) - if ≤50 bpm and decrease from baseline of ≥15 beats per minute (bpm); systolic blood pressure (SBP) - if ≤90 mm Hg and decrease from baseline of ≥20 mm Hg; diastolic blood pressure (DBP) - if ≤50 mm Hg and decrease from baseline of ≥15 mm Hg.
  Markedly abnormal increases: HR - if ≥110 bpm and increase from baseline of ≥15 bpm; SBP - if ≥180 mm Hg and increase from baseline of ≥20 mm Hg; DBP - if ≥105 mm Hg and increase from baseline of ≥15 mm Hg.
Time Frame: Post-baseline (at Week 4, 12, 20, 28, and 40 or endpoint)
Measure: Number; unit: Participants
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Number analyzed (Participants) | 32 | 79 | 107
Participants | 2 | 12 | 11

9. Primary Outcome: Number of Participants With Laboratory Values Outside Normal Range
Description: Normal ranges were provided by the central laboratory.
  Biochemistry = electrolytes, creatine kinase, liver enzymes, blood urea nitrogen, creatinine, alkaline phosphatase, protein, albumin
  Metabolic chemistry = cholesterol, glucose, triglycerides, glycosylated hemoglobin
  Endocrinology/miscellaneous = insulin, prolactin
  Hematology = hemoglobin, red blood cell count, white blood cell count, platelets, hematocrit, neutrophils, lymphocytes, monocytes, eosinophils, basophils
Time Frame: Week 40 or endpoint
Population: Number at risk = participants with either normal or abnormal baseline value and a non-missing value at endpoint.
  Actual at risk: 20-32 for placebo/asenapine arm; 50-78 for asenapine arm; 63-106 in olanzapine arm.
Measure: Number; unit: Participants
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Number analyzed (Participants) | 32 | 79 | 107
Participants
  Biochemistry | 25 | 76 | 115
  Metabolic chemistry | 17 | 32 | 96
  Endocrinology/miscellaneous | 7 | 35 | 39
  Hematology | 22 | 90 | 83

ADVERSE EVENTS:
Arm/Group | Placebo/Asenapine | Asenapine | Olanzapine
Serious Adverse Events (participants affected / at risk) | 2/32 | 6/79 | 9/107
Other Adverse Events (participants affected / at risk) | 12/32 | 28/79 | 34/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Asenapine (N=32) | Asenapine (N=79) | Olanzapine (N=107)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Death neonatal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Asenapine (N=32) | Asenapine (N=79) | Olanzapine (N=107)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 7 (7)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 6 (6)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 4 (6)
Weight decreased (Investigations) | 3 (3) | 4 (4) | 0 (0)
Weight increased (Investigations) | 1 (2) | 5 (5) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Parkinsonism (Nervous system disorders) | 2 (2) | 2 (2) | 1 (4)
Sedation (Nervous system disorders) | 1 (1) | 5 (5) | 5 (7)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 7 (8) | 5 (5)
Insomnia (Nervous system disorders) | 2 (5) | 6 (7) | 7 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If study is part of a multicenter trial, Investigator agrees that the first publication is to be a joint publication covering all centers. However, if a joint manuscript has not been submitted for publication within 12 mos of completion or termination of study at all participating sites, Investigator is free to publish separately.

The sponsor should review any publication prior to submission for publication to ensure no confidential information is released inadvertently.